CLINICAL TRIAL: NCT06125795
Title: Non-interventional Prospective Descriptive Study to Assess the Impact on Patient´s Well-being of Fixed-time Duration (FTD) and Continuous Oral Regimens for Newly Diagnosed and Relapsed/Refractory (R/R) Chronic Lymphocytic Leukemia (CLL) in Routine Clinical Practice in Spain
Brief Title: A Study to Assess Change in Functioning and Health Related Quality of Life in Adult Participants With Chronic Lymphocytic Leukemia (CLL) Receiving Oral Treatments in Routine Clinical Practice in Spain
Acronym: PROVIDENCE
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-280
Record Dates: First submitted 2023-10-24; First posted 2023-11-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Bruton Tyrosine Kinase Inhibitor; Patient-Reported Outcomes Measure; Patient-Reported Experience Measure; Venetoclax; Venclexta; Venclyxto; ABT-199; Patient Preferences; Cancer; PROVIDENCE
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Patient Preference; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic Lymphocytic Leukemia (CLL) Participants: Participants will receive oral treatments for CLL in accordance with approved local label.

SUMMARY:
Chronic lymphocytic leukemia (CLL) is the most common leukemia in the Western world. Since in most cases CLL remains an incurable disease, the goals of therapy are to improve quality of life and to prolong survival. This study will evaluate the participant's related outcomes and experience of CLL in adult participants who are treated in the Spain.

Study participants will receive oral treatments for CLL as prescribed by their study doctor in accordance with approved local label. Adult participants prescribed various treatments will be enrolled. Around 132 participants will be enrolled in the study in sites in Spain.

Participants will receive oral treatments for CLL according to the approved local label. The overall study duration will be 18 months.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Have documented chronic lymphocytic leukemia (CLL) according to International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria.
* Under oral treatment for CLL, either first-line or relapsed/refractory (R/R) therapy.
* Treatment for CLL started 9 months (+/- 4 weeks) before inclusion for first-line therapy or 21 months (+/- 4 weeks) before inclusion for R/R, under authorized conditions.
* In the opinion of the investigator, cognitive ability to understand and answer the questionnaires specified in the study protocol.
* Able to comply with the study protocol in the investigator's judgment.

Exclusion Criteria:

* Currently receiving any chemotherapy or chemoimmunotherapy.
* Transformation of CLL to aggressive non-Hodgkin's lymphoma (NHL) (Richter's transformation or pro-lymphocytic leukaemia).
* Currently participating in interventional research (not including non-interventional study, post-marketing observational study, or registry participation).
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with chronic lymphocytic leukemia (CLL) treated with fixed-time duration (FTD) or continuous oral regimens who attend to a regular follow up visit at a Spanish participating hospital will be eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Participant Functioning Measured Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) with the EORTC Chronic Lymphocytic Leukemia 17 (EORTC-CLL17) Supplement | Up to 27 Months
  The EORTC-CLL17 is a specific questionnaire that supplements the EORTC QLQ-C30 for participants with CLL.
  EORTC-CLL17 comprises 17 items divided into three subscales: symptom burden, physical condition/fatigue, and worries/fears about the health and functioning. The scores of each subscale are calculated based on the EORTC's protocol and then transformed to a 0 to 100 scale. A high score represents a high level of symptomology high level of physical condition/fatigue, and a high level of worries/fears about the health and functioning.
  EORTC QLQ-C30 is a questionnaire to assess the quality of life (QoL) of cancer participants. It is composed of five functional scales, three symptom scales, a global health status/QoL scale, and six single items. A high score represents high level of functioning, or QoL, but a high level of symptomology/problems.
Change in Participant Health-related Quality of Life (HRQoL)Measured Using the EORTC QLQ-C30 with the EORTC-CLL17 Supplement | Up to 27 Months
  The EORTC-CLL17 is a specific questionnaire that supplements the EORTC QLQ-C30 for participants with CLL.
  EORTC-CLL17 comprises 17 items divided into three subscales: symptom burden, physical condition/fatigue, and worries/fears about the health and functioning. The scores of each subscale are calculated based on the EORTC's protocol and then transformed to a 0 to 100 scale. A high score represents a high level of symptomology high level of physical condition/fatigue, and a high level of worries/fears about the health and functioning.
  EORTC QLQ-C30 is a questionnaire to assess the QoL of cancer participants. It is composed of five functional scales, three symptom scales, a global health status/QoL scale, and six single items. A high score represents a high level of functioning, or QoL, but a high level of symptomology/problems.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (25):
- Spain (25):
  - HUA - Txagorritxu /ID# 258263, Vitoria-Gasteiz, Alava
  - Sant Joan de Deu de Manresa /ID# 258266, Manresa, Barcelona
  - Hospital Universitari Mútua Terrassa /ID# 258267, Terrassa, Barcelona
  - Hospital Jerez De La Frontera /ID# 258282, Jerez de la Frontera, Cadiz
  - Hospital Comarcal de Laredo /ID# 258262, Laredo, Cantabria
  - Hospital Universitario Marques de Valdecilla /ID# 258261, Santander, Cantabria
  - Hospital Universitario Reina Sofia /ID# 271507, Córdoba, Cordoba
  - Hospital Universitario Dr. Negrin /ID# 258285, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario de León /ID# 271526, León, Leon
  - Hospital Universitario de Fuenlabrada /ID# 258275, Fuenlabrada, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca /ID# 262173, El Palmar, Murcia
  - Hospital Meixoeiro (CHUVI) /ID# 258286, Vigo, Pontevedra
  - Hospital de Cabueñes /ID# 263307, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias /ID# 271508, Oviedo, Principality of Asturias
  - Hospital Universitario de Galdakao /ID# 258264, Galdakao, Vizcaya
  - Hospital de Sant Joan Despi Moises Broggi /ID# 262284, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 258280, Granada
  - Hospital Lucus Augusti /ID# 271542, Lugo
  - Hospital Universitario de La Princesa /ID# 271506, Madrid
  - Hospital General Universitario Gregorio Maranon /ID# 258273, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 258269, Madrid
  - Hospital Universitario 12 de Octubre /ID# 258271, Madrid
  - Hospital Universitario La Paz /ID# 258270, Madrid
  - Hospital General Universitario Morales Meseguer /ID# 258284, Murcia
  - Hospital Universitario Virgen Macarena /ID# 258279, Seville

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-280